CLINICAL TRIAL: NCT00768300
Title: ARTEMIS-IPF: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multi-Center, Parallel-Group, Event Driven Study to Evaluate the Efficacy and Safety of Ambrisentan in Subjects With Early Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: (ARTEMIS-IPF) Randomized, Placebo-Controlled Study to Evaluate Safety and Effectiveness of Ambrisentan in IPF
Acronym: ARTEMIS-IPF
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-231-0101
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Results first posted 2014-04-08 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-02

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: idiopathic pulmonary fibrosis; interstitial lung disease; ambrisentan
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Lung Diseases, Interstitial | interventions — ambrisentan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ambrisentan (Experimental)
  Interventions: Drug: Ambrisentan
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ambrisentan — Ambrisentan (5mg or 10 mg tablet) was administered orally once daily.
  Other Names: Letairis®
  Arms: Ambrisentan
Drug: Placebo — Placebo to match ambrisentan was administered orally once daily.
  Arms: Placebo

SUMMARY:
The ARTEMIS-IPF study was conducted to determine if ambrisentan was effective in delaying disease progression and death in participants with idiopathic pulmonary fibrosis (IPF), to evaluate its safety, and to evaluate its effect on development of pulmonary hypertension, quality of life, and dyspnea (shortness of breath) symptoms in this participant population. Participants were randomized in a 2:1 ratio to receive ambrisentan or placebo, respectively. Participation in the study was to be up to 4 years, depending on how long it would take to enroll participants and observe study events. After randomization, visits to the clinic took place every 3 months, and laboratory procedures were performed every month.

ELIGIBILITY:
Inclusion Criteria:

* Male or females from 40 to 80 years of age
* Diagnosis of IPF
* Honeycombing (fibrosis in the lung) on high-resolution computerised tomography (HRCT) scan of less than or equal to 5%
* Willing and able to have 2 right heart catheterizations performed
* Willing to have monthly lab tests to monitor liver function
* Able to perform the 6 minute walk test (indicated adequate physical function)
* Must have meet lung function requirements
* Normal liver function tests
* Negative serum pregnancy test
* Willing to use at least 2 reliable methods of contraception
* Able to understand and willing to sign informed consent form

Exclusion Criteria:

* No restrictive lung disease (other than usual interstitial pneumonia or IPF)
* No obstructive lung disease
* No recent or active respiratory exacerbations
* No recent hospitalization for an IPF exacerbation
* No recent history of alcohol abuse
* Chronic sildenafil (or same drug class) use for pulmonary hypertension
* Chronic treatment with certain medications for IPF within 30 days of randomization
* No other serious medical conditions

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Actual)
Dates: Start 2008-12; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ganesh Raghu, MD, Study Chair — University of Washington, Div. of Pulmonary and Critical Care Medicine Chair
Locations (168):
- United States (55):
  - University of Alabama at Birmingham Hospital, Birmingham, Alabama
  - Pulmonary Associates, Phoenix, Arizona
  - Scottsdale, Arizona
  - David Geffen School of Medicine at UCLA(Harbor-UCLA Medical Center), Los Angeles, California
  - University of California, Davis, Sacramento, California
  - San Diego, California
  - San Francisco, California
  - Stanford University, Stanford, California
  - National Jewish Medical And Research Center, Denver, Colorado
  - Newark, Delaware
  - Bay Area Chest Physicians, Clearwater, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Tampa, Florida
  - Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Council Bluffs, Iowa
  - Kentuckiana Pulmonary Association, Louisville, Kentucky
  - Louisville, Kentucky
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Saint Lukes Foundation, Chesterfield, Missouri
  - Dartmouth Medical School, Lebanon, New Hampshire
  - New Brunswick, New Jersey
  - Piscataway, New Jersey
  - Pulmonary & Allergy Associates, Summit, New Jersey
  - Pulmonary And Critical Care Services, P.C., Albany, New York
  - Winthrop University Hospital, Mineola, New York
  - New Hyde Park, New York
  - New York, New York
  - Columbia University Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Columbus, Ohio
  - The Oregon Clinic, P.C., Portland, Oregon
  - University of Pennsylvania Health Systems, Philadelphia, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - The Reading Hospital and Medical Center, Reading, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Lexington, South Carolina
  - Spartanburg, South Carolina
  - Nashville, Tennessee
  - Houston, Texas
  - McKinney, Texas
  - Provo, Utah
  - Salt Lake City, Utah
  - Charlottesville, Virginia
  - Falls Church, Virginia
  - Lynchburg, Virginia
  - Everett, Washington
  - Seattle, Washington
- Argentina (4):
  - Mar del Plata, Buenos Aires
  - Buenos Aires
  - Mar Del Plata, Buenos Aires
  - San Miguel de Tucumán
- Australia (8):
  - Concord, New South Wales
  - Darlinghurst, New South Wales
  - Chermside, Queensland
  - Woodville, South Australia
  - Hobart, Tasmania
  - Parkville, Victoria
  - Prahran, Victoria
  - Perth, Western Australia
- Austria (4):
  - Graz
  - Innsbruck
  - Linz
  - Vienna
- Belgium (4):
  - Anderlecht
  - Brussels
  - Leuven
  - Yvoir
- Brazil (7):
  - São Paulo, São Paulo
  - Belo Horizonte
  - Florianópolis
  - Goiânia
  - Porto Alegre
  - Rio de Janeiro
  - Santo André
- Canada (7):
  - Calgary, Alberta
  - Edmondton, Alberta
  - Vancouver, British Columbia
  - St. John's, Newfoundland and Labrador
  - Montreal, Quebec
  - Sainte-Foy, Quebec
  - Toronto
- Chile (3):
  - Santiago
  - Talcahuano
  - Valparaíso
- Colombia (2):
  - Bogotá
  - Floridablanca
- Czechia (6):
  - Brno
  - Hradec Králové
  - Jihlava
  - Liberec
  - Olomouc
  - Pilsen
- France (8):
  - Lille
  - Marseille
  - Montpellier
  - Nice
  - Paris
  - Pessac
  - Rennes
  - Tours
- Germany (9):
  - Berlin
  - Coswig
  - Donaustauf
  - Essen
  - Freiburg im Breisgau
  - Greifswald
  - Heidelberg
  - Löwenstein
  - München
- Dublin, Ireland
- Israel (8):
  - Ashkelon
  - Beersheba
  - Haifa
  - Jerusalem
  - Petah Tikva
  - Rehovot
  - Tel Aviv
  - Tel Litwinsky
- Italy (10):
  - Catania
  - Forlì
  - Milan
  - Modena
  - Napoli
  - Padua
  - Palermo
  - Roma
  - Siena
  - Torino
- Mexico (6):
  - Guadalajara, Jalisco
  - Monterrey, Nuevo León
  - Huixquilucan Edo. de Mexico
  - Mexico City, DF
  - Monterrey
  - Zapopan, Jalisco
- Almelo, Netherlands
- Peru (2):
  - Callao
  - Lima
- Poland (2):
  - Bydgoszcz
  - Lodz
- Spain (9):
  - Cadiz, Andalusia
  - Hospital Virgen del Rocio, Seville, Andalusia
  - Complejo Asistencial Universitario de León, León, Castilla
  - Pontevedra, Galicia
  - Pozuelo de Alarcón, Madrid, Communidad de
  - Oviedo, Principality of Asturias
  - Badalona
  - Barcelona
  - Madrid
- Switzerland (3):
  - Basel
  - Bern
  - Lausanne
- United Kingdom (9):
  - Sheffield, South Yorkshire
  - Chertsey, Surrey
  - Cambridge
  - Chelmsford
  - Edinburgh
  - Glasgow
  - Liverpool
  - London
  - Mancesheter

REFERENCES:
- [Result] Raghu G, Behr J, Brown KK, Egan JJ, Kawut SM, Flaherty KR, Martinez FJ, Nathan SD, Wells AU, Collard HR, Costabel U, Richeldi L, de Andrade J, Khalil N, Morrison LD, Lederer DJ, Shao L, Li X, Pedersen PS, Montgomery AB, Chien JW, O'Riordan TG; ARTEMIS-IPF Investigators*. Treatment of idiopathic pulmonary fibrosis with ambrisentan: a parallel, randomized trial. Ann Intern Med. 2013 May 7;158(9):641-9. doi: 10.7326/0003-4819-158-9-201305070-00003. PMID 23648946
- [Derived] Raghu G, Lynch D, Godwin JD, Webb R, Colby TV, Leslie KO, Behr J, Brown KK, Egan JJ, Flaherty KR, Martinez FJ, Wells AU, Shao L, Zhou H, Pedersen PS, Sood R, Montgomery AB, O'Riordan TG. Diagnosis of idiopathic pulmonary fibrosis with high-resolution CT in patients with little or no radiological evidence of honeycombing: secondary analysis of a randomised, controlled trial. Lancet Respir Med. 2014 Apr;2(4):277-84. doi: 10.1016/S2213-2600(14)70011-6. Epub 2014 Feb 18. PMID 24717624
- [Derived] Chien JW, Richards TJ, Gibson KF, Zhang Y, Lindell KO, Shao L, Lyman SK, Adamkewicz JI, Smith V, Kaminski N, O'Riordan T. Serum lysyl oxidase-like 2 levels and idiopathic pulmonary fibrosis disease progression. Eur Respir J. 2014 May;43(5):1430-8. doi: 10.1183/09031936.00141013. Epub 2013 Oct 31. PMID 24177001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in a total of 136 study sites in North and South America, Europe, and Australia. The first participant was screened on 10 December 2008. The last participant observation was on 28 February 2011.
Pre-assignment Details: 494 participants were randomized; 492 participants were treated, and comprise the Safety Analysis Set and the Full Analysis Set.
Groups:
- Ambrisentan: Ambrisentan (5 mg or 10 mg tablet) administered orally once daily
- Placebo: Placebo to match ambrisentan administered orally once daily
Period: Overall Study
Arm/Group | Ambrisentan | Placebo
Started | 330 | 164
Randomized and Treated | 329 | 163
Completed | 1 | 1
Not Completed | 329 | 163
Not completed — Randomized but not treated | 1 | 1
Not completed — Adverse Event | 10 | 2
Not completed — Protocol Violation | 6 | 1
Not completed — Withdrawal by Subject | 13 | 7
Not completed — Physician Decision | 2 | 3
Not completed — Study discontinued by Sponsor | 271 | 140
Not completed — Death | 21 | 5
Not completed — Subject moved to pursue lung transplant | 1 | 1
Not completed — Screen failure following randomization | 1 | 0
Not completed — Received lung transplant | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Began prohibited concomitant medication | 0 | 1
Not completed — Treated but never dosed with Study drug | 1 | 0
Not completed — Missing data | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: participants who were randomized and treated
Groups:
- Total: Total of all reporting groups
Arm/Group | Ambrisentan | Placebo | Total
Number analyzed (Participants) | 329 | 163 | 492
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (7.4) | 66.1 (7.1) | 65.9 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 52 | 137
  Male | 244 | 111 | 355
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African Heritage | 1 | 0 | 1
  White | 293 | 145 | 438
  Asian | 4 | 1 | 5
  American Indian or Alaskan Native | 1 | 1 | 2
  Other | 27 | 16 | 43
  Not Permitted | 3 | 0 | 3
Region of Enrollment [Number; unit: participants] — All participants who were randomized are presented in Region of Enrollment (ambrisentan = 330; placebo = 164)
  participants
    United States | 141 | 62 | 203
    Canada | 25 | 14 | 39
    Australia | 22 | 12 | 34
    France | 21 | 10 | 31
    Germany | 17 | 9 | 26
    Brazil | 18 | 6 | 24
    Peru | 12 | 6 | 18
    Czech Republic | 10 | 6 | 16
    Israel | 8 | 7 | 15
    Italy | 11 | 3 | 14
    Belgium | 7 | 6 | 13
    Colombia | 8 | 3 | 11
    Mexico | 5 | 4 | 9
    United Kingdom | 3 | 6 | 9
    Spain | 7 | 1 | 8
    Poland | 3 | 3 | 6
    Switzerland | 5 | 1 | 6
    Austria | 2 | 2 | 4
    Chile | 3 | 1 | 4
    Argentina | 1 | 2 | 3
    Ireland | 1 | 0 | 1
Baseline Pulmonary Hypertension (PH) per interactive voice response system (IVRS) [Number; unit: participants]
  No | 293 | 145 | 438
  Yes | 36 | 18 | 54
Smoking status [Number; unit: participants] — Smoking status data is missing for one participant randomized to placebo.
  participants
    Never | 105 | 53 | 158
    Current | 7 | 5 | 12
    Former | 217 | 104 | 321
Surgical lung biopsy (SLB) to Confirm Diagnosis of IPF (per IVRS) [Number; unit: participants]
  No | 175 | 87 | 262
  Yes | 154 | 76 | 230
Disease duration [Mean (Standard Deviation); unit: years] | 1.13 (1.39) | 0.91 (1.19) | 1.06 (1.33)
Forced vital capacity (FVC) percent predicted [Least Squares Mean (Standard Deviation); unit: percentage of FVC % predicted] | 68.74 (13.12) | 69.86 (13.75) | 69.11 (13.33)
Six mile walk test (6MWT) [Mean (Standard Deviation); unit: meters] | 410.4 (118.7) | 420.5 (121.4) | 413.7 (119.6)
Hemoglobin Adjusted Diffusing lung capacity for carbon monoxide (DLCO) percent predicted [Least Squares Mean (Standard Deviation); unit: percentage of DLCO % predicted] | 42.04 (13.77) | 45.57 (13.25) | 43.20 (13.69)
Prior IPF Medications [Number; unit: participants] — Prior IPF Medications data is missing for one participant randomized to placebo.
  participants
    No | 205 | 97 | 302
    Yes | 124 | 65 | 189
N-acetylcysteine (NAC) Use [Number; unit: participants] — NAC is a therapy commonly used in the treatment of IPF. NAC use data is missing for two participants randomized to placebo.
  participants
    No | 310 | 153 | 463
    Yes | 19 | 8 | 27

OUTCOME MEASURES:

1. Primary Outcome: Time to Death or Disease (IPF) Progression.
Description: The median time to death or disease progression was based on Kaplan-Meier (KM) estimates of pooling over strata, and was defined as the first occurrence of any of the following:
  * Either 1) a decrease of ≥ 10% in FVC (L) and a decrease of ≥ 5% in diffuse lung capacity for carbon monoxide (DLCO) (ml/min/mmHg), or 2) a decrease of ≥ 5% in FVC (L) and a decrease of ≥ 15% in DLCO (ml/min/mmHg); deterioration in FVC and DLCO must be confirmed at the subsequent visit within 28 (± 14) days
  * Respiratory hospitalization (hospitalization involving worsening of, or deterioration in respiratory symptoms, gas exchange/hypoxemia, or radiographic findings on chest x-ray or high-resolution computerised tomography (HRCT) scan
  * All-cause mortality
Time Frame: Up to 48 months
Population: Full Analysis Set: participants who were randomized and treated
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Ambrisentan | Placebo
Number analyzed (Participants) | 329 | 163
weeks | 84.14 [36.00 to NA] — Insufficient data for estimation due to study termination | NA [60.00 to NA] — Insufficient data for estimation due to study termination
Statistical Analysis 1: Comparison: Ambrisentan vs Placebo; Test type: Superiority or Other; p = 0.010, Log Rank — P-value was based on a stratified log-rank test with strata of baseline presence of pulmonary hypertension and whether a surgical lung biopsy was performed with definite or probable usual interstitial pneumonia (UIP) based on core pathology review; Hazard Ratio (HR) = 1.74, 95% CI 2-sided [1.14 to 2.66] — The hazard ratio was based on a stratified Cox proportional hazards model with strata of baseline presence of pulmonary hypertension and whether a surgical lung biopsy was performed with definite or probable UIP based on core pathology review

2. Secondary Outcome: Proportion of Participants With No Disease Progression or Death at 48 Weeks
Description: The proportion of participants with no disease progression or death is presented as a percentage using a Kaplan-Meier (KM) estimate of survival or not experiencing disease progression.
Time Frame: Baseline and Week 48
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Ambrisentan | Placebo
Number analyzed (Participants) | 329 | 163
percentage of participants | 65 | 80

3. Secondary Outcome: Change in FVC % Predicted at Week 48
Description: FVC is defined as the volume of air (liters) that can forcibly be blown out after taking a full breath. FVC % predicted is defined as FVC % of the participant divided by the average FVC % in the population for any person of similar age, sex, and body composition.
Time Frame: Baseline and Week 48
Population: Participants in the Full Analysis Set with evaluable change data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change in FVC % predicted
Arm/Group | Ambrisentan | Placebo
Number analyzed (Participants) | 163 | 80
percent change in FVC % predicted | -10.24 (25.95) | -5.28 (15.68)
Statistical Analysis 1: Comparison: Ambrisentan vs Placebo; Test type: Superiority or Other; p = 0.086, Van Elteren test — P-value was calculated using the Van Elteren test with strata of baseline presence of PH and whether a SLB was performed with definite or probable UIP based on core pathology review; Point estimate = 4.29, 95% CI 2-sided [-0.805 to 9.376] — The point estimate and 95% confidence interval (CI) were based on the Hodges-Lehmann Estimate of treatment effect for percent change from baseline

4. Secondary Outcome: Change in DLCO % Predicted at Week 48
Description: DLCO is the extent to which oxygen passes from the air sacs of the lungs into the blood. DLCO % predicted is defined as DLCO % of the participant divided by the average DLCO % in the population for any person of similar age, sex and body composition.
Time Frame: Baseline and Week 48
Population: Participants in the Full Analysis Set with evaluable change data were analyzed.
Measure: Mean (Standard Deviation); unit: percent change in DLCO % predicted
Arm/Group | Ambrisentan | Placebo
Number analyzed (Participants) | 163 | 80
percent change in DLCO % predicted | -2.68 (27.60) | -11.28 (32.06)
Statistical Analysis 1: Comparison: Ambrisentan vs Placebo; Test type: Superiority or Other; p = 0.250, Van Elteren test — [p-value comment as in outcome 3, analysis 1]; Point estimate = 2.85, 95% CI 2-sided [-2.20 to 7.90] — The point estimate and its 95% CI were based on the Hodges-Lehmann Estimate of treatment effect for percent change from baseline

5. Secondary Outcome: Change in 6MWT at Week 48
Description: The 6MWT is a measure of exercise tolerance, and measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface.
Time Frame: Baseline and Week 48
Population: Participants in the Full Analysis Set with evaluable change data were analyzed.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Ambrisentan | Placebo
Number analyzed (Participants) | 162 | 80
meters | -52.5 (148.7) | -10.6 (89.8)
Statistical Analysis 1: Comparison: Ambrisentan vs Placebo; Test type: Superiority or Other; p = 0.150, Van Elteren test — [p-value comment as in outcome 3, analysis 1]; Point estimate = 16.00, 95% CI 2-sided [-5.00 to 37.00] — The point estimate and 95% CI were based on the Hodges-Lehmann Estimate of treatment effect for percent change from baseline

6. Secondary Outcome: Change in Quality of Life (QOL) Score at Week 48 as Assessed by the Short-Form 36® (SF-36)
Description: The range of each health domain score is 0-100, with 0 indicating a poorer health state and 100 indicating a better health state. An increase in score indicates an improvement in health state.
Time Frame: Baseline and Week 48
Population: Participants in the Full Analysis Set with evaluable change data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ambrisentan | Placebo
Number analyzed (Participants) | 158 | 78
units on a scale
  Physical function | -1.65 (10.86) | -2.60 (7.25)
  General Health | -2.81 (9.77) | -1.95 (8.63)
  Vitality | -1.67 (12.67) | -0.12 (7.69)

7. Secondary Outcome: Change in Quality of Life (QOL) Score at Week 48 as Assessed by the St. George's Respiratory Questionnaire (SGRQ)
Description: The SGRQ is designed to measure impact on overall health, daily life, and perceived well-being in participants with obstructive airways disease. The range of each score is 0-100, with 0 indicating fewer limitations and 100 indicating more limitations; an increase in score indicates an increase in limitations.
Time Frame: Baseline and Week 48
Population: Participants in the Full Analysis Set with evaluable change data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ambrisentan | Placebo
Number analyzed (Participants) | 159 | 78
units on a scale
  Symptoms Score | 3.30 (22.11) | 2.84 (20.43)
  Activity Score | 5.54 (19.38) | 2.05 (16.47)
  Impacts Score | 4.68 (24.07) | 3.09 (15.80)
  Total Score | 4.70 (19.92) | 3.04 (13.80)

8. Secondary Outcome: Change in Dyspnea Score at Week 48 as Assessed by the Transitional Dyspnea Index (TDI)
Description: The transitional focal score (-9 to 9) is the sum of relative change from baseline for the Functional Impairment, Magnitude of Task, and Magnitude of Effort scores (each -3 to 3 scale). A TDI score of -9 represents a maximum degradation of all three tests; a score of 9 represents a maximum improvement of all three tests.
Time Frame: Baseline and Week 48
Population: Participants in the Full Analysis Set with evaluable change data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ambrisentan | Placebo
Number analyzed (Participants) | 163 | 80
units on a scale | -1.23 (3.74) | -0.84 (2.99)
Statistical Analysis 1: Comparison: Ambrisentan vs Placebo; Test type: Superiority or Other; p = 0.793, Wilcoxon (Mann-Whitney) — The p-value was based on a Wilcoxon rank sum test stratified by baseline pulmonary hypertension (Yes/No) and surgical lung biopsy was performed with definite or probable UIP based on core pathology review (Yes/No); Point estimate = 0.50, 95% CI 2-sided [0.00 to 1.00] — The point estimate and 95% confidence interval were based on the Hodges-Lehmann Estimate of treatment effect

9. Secondary Outcome: Percentage of Participants Who Developed PH on Study
Description: The percentage of participants known to have developed pulmonary hypertension on study documented by right heart catheterization (RHC) was analyzed. RHC was done at baseline and 48 weeks, or at the early termination visit.
Time Frame: Up to 48 weeks
Population: Participants in the Full Analysis Set without PH at baseline were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Ambrisentan | Placebo
Number analyzed (Participants) | 293 | 145
percentage of participants | 0.7 | 2.1

ADVERSE EVENTS:
Time Frame: Up to 48 months
Arm/Group | Ambrisentan | Placebo
Serious Adverse Events (participants affected / at risk) | 73/329 | 25/163
Other Adverse Events (participants affected / at risk) | 227/329 | 104/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ambrisentan (N=329) | Placebo (N=163)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 3 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 4 | 0
Cardiomegaly (Cardiac disorders) | 1 | 0
Dilatation atrial (Cardiac disorders) | 1 | 0
Tricuspid valve incompetence (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Extrasystoles (Cardiac disorders) | 1 | 0
Electromechanical dissociation (Cardiac disorders) | 1 | 0
Acute vestibular syndrome (Ear and labyrinth disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Choroidal haemorrage (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 4 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Colitis (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Colonic polyp (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Aptyalism (Gastrointestinal disorders) | 0 | 1
Oedema peripheral (General disorders) | 4 | 1
Oedema (General disorders) | 1 | 0
Chest pain (General disorders) | 2 | 1
Pain (General disorders) | 2 | 0
Pyrexia (General disorders) | 2 | 0
Fatigue (General disorders) | 2 | 0
Catheter site haemorrhage (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 0
Hyperthermia (General disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 9 | 2
Bronchitis (Infections and infestations) | 3 | 0
Lobar pneumonia (Infections and infestations) | 1 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 2 | 1
Infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0
Endocarditis bacterial (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 2 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Conjunctivitis viral (Infections and infestations) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
Electrocardiogram ST-T segment abnormal (Investigations) | 1 | 0
Electrocardiogram T wave inversion (Investigations) | 1 | 0
Computerised tomogram thorax abnormal (Investigations) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1
Clubbing (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Headache (Nervous system disorders) | 5 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Somnolence (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Coma (Nervous system disorders) | 1 | 0
Grand mal convulsion (Nervous system disorders) | 1 | 0
Nerve compression (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 3 | 0
Delirium (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 2 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 20 | 4
Emphysema (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 | 2
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 4 | 1
Hypertension (Vascular disorders) | 3 | 0
Subclavian vein thrombosis (Vascular disorders) | 1 | 0
Flushing (Vascular disorders) | 1 | 0
Hot flush (Vascular disorders) | 1 | 0
Cardiac ventricular disorder (Cardiac disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ambrisentan (N=329) | Placebo (N=163)
Oedema peripheral (General disorders) | 73 | 14
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 47 | 18
Headache (Nervous system disorders) | 47 | 17
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 40 | 11
Nasopharyngitis (Infections and infestations) | 37 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 34 | 20
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 19 | 2
Bronchitis (Infections and infestations) | 23 | 15
Fatigue (General disorders) | 22 | 14
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 27 | 6
Constipation (Gastrointestinal disorders) | 19 | 10
Diarrhoea (Gastrointestinal disorders) | 20 | 8
Sinusitis (Infections and infestations) | 20 | 6
Respiratory tract infection (Infections and infestations) | 9 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 18 | 5
Dizziness (Nervous system disorders) | 20 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 8 | 9
Nausea (Gastrointestinal disorders) | 15 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years